CLINICAL TRIAL: NCT00002762
Title: MENSTRUAL CYCLE AND SURGICAL TREATMENT OF BREAST CANCER
Brief Title: Correlation of Menstrual Cycle Phase at Time of Primary Surgery With 5-Year Disease-Free Survival in Women With Stage I or Stage II Breast Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Other Study IDs: NCCTG-N9431; NCI-2012-02243 (Registry Identifier: CTRP (Clinical Trials Reporting System)); NSABP-BI-65; CDR0000064717 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Perioperative/Postoperative Complications
Keywords: stage I breast cancer; stage II breast cancer; perioperative/postoperative complications
MeSH Terms: conditions — Breast Neoplasms; Postoperative Complications | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patient interviewing + blood sampling: Patients were interviewed at the time of the primary cancer surgery to determine the menstrual history. Blood sampling occurred within 1 day of surgery, and serum samples were shipped frozen to a central laboratory (Mayo Medical Laboratory, Rochester, MN) for E2, Pg, and LH determinations. Serum hormone levels, menstrual cycle length, and day of last menses were used to determine the menstrual phase at which surgery occurred.
  Patients were observed every 6 months for the first year postregistration and annually for the next 2 to 10 years postregistration for adjuvant therapy information, disease recurrence, and death.
  Interventions: Behavioral: patient interviewing to obtain menstrual history; Procedure: blood sampling

INTERVENTIONS:
Behavioral: patient interviewing to obtain menstrual history
Procedure: blood sampling

SUMMARY:
RATIONALE: Timing of breast cancer surgery may improve effectiveness of treatment and may help patients live longer.

PURPOSE: Clinical trial to determine whether timing of primary surgery in relation to menstrual cycle is associated with disease-free survival 5 years after surgery in women who have stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Document menstrual phase (follicular vs luteal) by circulating hormones and menstrual history at the time of primary surgery in premenopausal women with stage I or II breast cancer.
* Correlate menstrual phase at primary surgery with 5-year disease-free survival in these patients.
* Compare the menstrual cycle data obtained by hormone levels and study-specific menstrual cycle history with information recorded in the general written record.
* Compare the menstrual cycle data (e.g., hormone levels and cycle history) for these women with the data for the general population.
* Estimate the disease-free survival of women who undergo a 2-stage surgical procedure with cancer found at both stages when the surgery is not confined to the same menstrual cycle phase.

Premenopausal women age 18 to 55 years, who were interviewed for menstrual history and who were surgically treated for stages I to II breast cancer, had serum drawn within 1 day of surgery for estradiol, progesterone, and luteinizing hormone levels. Menstrual history and hormone levels were used to determine menstrual phase: luteal, follicular, and other. Disease-free survival (DFS) and overall survival (OS) rates were determined by Kaplan-Meier method and were compared by using the log-rank test and Cox proportional hazard modeling.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 18 to 55 years
2. Regular menstrual cycles of 21- to 35-days duration
3. Pathologic stages I to II breast cancer, in whom all gross disease-including ductal carcinoma in situ-was surgically removed either in a one-stage or two-stage procedure.
4. required serum be drawn within 1 calendar day of the lumpectomy/mastectomy for women who underwent a one-stage procedure and within 1 calendar day of each stage for women who underwent a two-stage procedure.

Exclusion Criteria:

1. Lactation within the past 3 months
2. galactorrhea
3. neoadjuvant therapy
4. previous breast cancer, and history of any cancer (except squamous or basal cell skin carcinoma) in which the patient was not disease-free for at least 10 years

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This trial enrolled premenopausal women age 18 to 55 years who had regular menstrual cycles of 21- to 35-days duration and pathologic stages I to II breast cancer, in whom all gross disease-including ductal carcinoma in situ-was surgically removed either in a one-stage or two-stage procedure.
Sampling Method: Non-Probability Sample
Enrollment: 1118 (Actual)
Dates: Start 1996-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
disease-free survival | Up to 5 years
overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clive S. Grant, MD, Study Chair — Mayo Clinic
Locations (54):
- United States (52):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Scripps Cancer Center at Scripps Clinic, La Jolla, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Hartford Hospital, Hartford, Connecticut
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - CCOP - Evanston, Evanston, Illinois
  - Rockford Clinic, Rockford, Illinois
  - Community Regional Cancer Care, Indianapolis, Indiana
  - CCOP - Wichita, Wichita, Kansas
  - Eastern Maine Medical Center, Bangor, Maine
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Warren Grant Magnuson Clinical Center, Bethesda, Maryland
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Akron City Hospital, Akron, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - South Pointe Hospital, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - St. Luke's Hospital and Health Network - Bethlehem, Bethlehem, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Wellspan Health - York Cancer Center, York, Pennsylvania
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Eastern Virginia Medical School, Norfolk, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Canada (2):
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Jewish General Hospital - Montreal, Montreal, Quebec

REFERENCES:
- [Result] Grant CS, Ingle JN, Suman VJ, Dumesic DA, Wickerham DL, Gelber RD, Flynn PJ, Weir LM, Intra M, Jones WO, Perez EA, Hartmann LC. Menstrual cycle and surgical treatment of breast cancer: findings from the NCCTG N9431 study. J Clin Oncol. 2009 Aug 1;27(22):3620-6. doi: 10.1200/JCO.2008.21.3603. Epub 2009 Jun 1. PMID 19487378